CLINICAL TRIAL: NCT07368205
Title: Preoperative Risk Stratification in Endometrial Cancer Using Expert Ultrasound and Molecular Classification for Tailoring Lymph Node Staging: Multicentric Prospective Observational Study
Brief Title: Preoperative Risk Stratification in Endometrial Cancer for Tailoring Lymph Node Staging
Acronym: PRSTEC_multipr
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Other Study IDs: 202511P08
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; molecular classification; expert ultrasonography; lymph node staging
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — preoperative biopsy specimen - endometrial tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
The goal of this observational study is to evaluaty the accuracy of current risk stratification of patients with endometrial cancer and to redefine lymph node staging recommendations based on real-world clinical data. The main question it aims to answer is:

Is there any group of patients who doesn't need lymph node staging for proper indication of adjuvant treatment? Participants are note taking any intervention. They are treated according to current standard of care and followed 3-years after primary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years with newly diagnosed endometrial cancer (any histology)
* Undergoing primary surgical management
* Preoperative expert ultrasound, CT scan (could be waived in low risk cases)
* Preoperatively early-stage (stage I-II) of EC
* SLN mapping attempted intraoperatively
* FFPE tumor tissue available for molecular and IHC testing from biopsy
* Signed informed consent with the participation in the study

Exclusion Criteria:

* Neoadjuvant treatment
* Recurrent or metastatic disease at diagnosis
* Inadequate imaging or tissue samples
* Cancer synchronous duplicity
* Prior oncological treatment within the last five years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologicaly confirmed endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
The accuracy of preoperative risk stratification | From enrollment to the first follow-up visit at 4 weeks after surgery.
Determination of specific groups for whom: 1) lymph node staging is crucial for changing risk category and adjuvant treatment decisions, and 2) lymph node staging could be safely omitted | From enrollment to the first follow-up visit at 4 weeks after surgery.

IPD SHARING:
Plan to Share IPD: Undecided